CLINICAL TRIAL: NCT02613923
Title: A Pilot Sleep Intervention to Improve Outcomes Among Women at High Risk of Breast Cancer
Brief Title: A Sleep Intervention to Improve Outcomes Among Women at High Risk of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASE6114
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Sleep
Keywords: Breast Cancer; GO! to sleep; sleep
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GO! To Sleep (Experimental): Participants in the intervention group will be provided with a code and website address to participate in this program. This program includes reminder emails and is 6 weeks in duration. Participants will be given a blood draw to measure biomarkers.
  Interventions: Behavioral: GO! To Sleep; Procedure: Blood Draw; Other: Pittsburgh Sleep Quality Index (PSQI); Other: Insomnia Severity Index (ISI); Other: SF-12 quality of life survey
- informational control (Active Comparator): Participants in the control group will receive weekly emails with sleep information and the health benefits of sleep for 6 weeks.Participants will be given a blood draw to measure biomarkers.
  Interventions: Behavioral: Sleep information; Procedure: Blood Draw; Other: Pittsburgh Sleep Quality Index (PSQI); Other: Insomnia Severity Index (ISI); Other: SF-12 quality of life survey

INTERVENTIONS:
Behavioral: GO! To Sleep — Controlled sleep intervention. Provide online education and reminder emails on improving sleep behavior
  Arms: GO! To Sleep
Behavioral: Sleep information — Participants will receive weekly emails on the health benefits of sleep for 6 weeks
  Arms: informational control
Procedure: Blood Draw — blood sample measured for stress and sleep markers
  Other Names: biomarker measurement
Other: Pittsburgh Sleep Quality Index (PSQI) — Assessment of sleep quality. This is a continuous measure from 0 (best) to 21 (worst). Sleep duration will be obtained directly from responses.
Other: Insomnia Severity Index (ISI)
Other: SF-12 quality of life survey

SUMMARY:
Participants are asked to participate in a research study of the effect of a sleep intervention on improving sleep habits and reducing their risk of breast cancer.

Participants are asked to participate in this research study because they have been identified as being at higher than average risk of developing breast cancer.

The purpose of this study is to compare women who get a sleep intervention to women who do not get a sleep intervention. This study team will compare these two groups of women to see if the sleep intervention improves their sleep and if it lowers markers of inflammation that have been associated with an increased risk of breast cancer.

DETAILED DESCRIPTION:
Objective 1: To test the effectiveness of the GO! To Sleep program at improving the sleep duration and sleep quality in women at high risk of breast cancer.

Objective 2: To test the effectiveness of improvements in sleep quality and/or duration due to the GO! To Sleep program on biomarkers of inflammation in women at high risk of breast cancer.

Objective 3: To evaluate the effectiveness of improvements in health-related quality of life after the GO! To Sleep in women at high risk of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women at high risk of breast cancer due to one or more of the following:

   * Carry deleterious mutations in the BRCA1, BRCA2, PTEN, TP53, STK11, or CDH1 genes
   * Previous diagnosis of lobular carcinoma in situ (LCIS), atypical ductal hyperplasia (ADH) or atypical lobular hyperplasia (ALH)
   * Lifetime risk of 20% or greater as calculated by the National Cancer Institute (NCI) Breast Cancer Risk Assessment Tool or the Tyrer-Cuzick IBIS Risk Assessment Tool
2. Ability to access the internet and watch videos online.
3. Valid email address.
4. Self-reported sleep duration of 6 hours per night or less

Exclusion Criteria:

1. Previous diagnosis of cancer.
2. Lack of ability to read and converse in English.
3. Lack of ability to give informed consent.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
Difference in Change in Pittsburgh Sleep Quality Index (PSQI) score between groups | Change from baseline to post intervention, around 8 weeks after baseline
  Sleep quality will be measured by the PSQI which is a continuous measure from 0 (best) to 21 (worst)
Difference in change in Insomnia Severity Index (ISI) score between groups | Change from baseline to post intervention, around 8 weeks after baseline
  Sleep quality will be measured with the insomnia severity index (ISI). A validated instrument for sleep quality
Difference in change in sleep duration between groups | Change from baseline to post intervention, around 8 weeks after baseline
  Sleep duration will be obtained by self-report from responses to the PSQI

SECONDARY OUTCOMES:
Difference in change of SF-12 score from baseline to post-intervention between groups | Change from baseline to 6 months post intervention
  The effectiveness of changing health-related quality of life after the GO! To Sleep program will he measured with the self-reported survey SF-12
Correlation of joint changes in biomarker levels with PSQI and ISI | Change from baseline to 6 months post intervention
  This study will correlate the joint changes in biomarker level with the changes in sleep quality and sleep duration
Difference in Change in Pittsburgh Sleep Quality Index (PSQI) score between groups | Change from baseline to 6 months post intervention
  Long term sleep quality will be measured by the PSQI which is a continuous measure from 0 (best) to 21 (worst)
Difference in change in Insomnia Severity Index (ISI) score between groups | Change from baseline to 6 months post intervention
  Sleep quality will be measured with the insomnia severity index (ISI). A validated instrument for sleep quality
Difference in change in sleep duration between groups | Change from baseline to 6 months post intervention
  Sleep duration will be obtained by self-report from responses to the PSQI

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Thompson, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States